CLINICAL TRIAL: NCT02953457
Title: A Phase I/II Evaluation of Olaparib in Combination With Durvalumab (Medi4736) and Tremelimumab in the Treatment of Recurrent Platinum Sensitive or Resistant or Refractory Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer in Patients Who Carry a BRCA1 or BRCA2 Mutation
Brief Title: Olaparib, Durvalumab, and Tremelimumab in Treating Patients With Recurrent or Refractory Ovarian, Fallopian Tube or Primary Peritoneal Cancer With BRCA1 or BRCA2 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 288216; NCI-2016-01598 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 288216 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation; Ovarian Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; olaparib; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib, tremelimumab, durvalumab) (Experimental): Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Drug: Olaparib; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Olaparib — Given PO
  Other Names: AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
This phase I/II trial studies the side effects and best dose of olaparib when give together with durvalumab and tremelimumab and to see how well they work in treating patients with ovarian, fallopian tube, or primary peritoneal cancer with BRCA1 or BRCA2 genetic mutation that has come back or has not responded to treatment. Drugs, such as olaparib, may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and kill tumors cells with BRCA1 or BRCA2 mutation. Monoclonal antibodies, such as durvalumab and tremelimumab, may help stimulate the immune system in different ways to attack and stop tumor cells from growing. Giving olaparib with durvalumab and tremelimumab may work better in treating patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and toxicity of the combination of PARP inhibitor olaparib with anti-PD-L1 antibody durvalumab and anti-CTLA4 antibody tremelimumab. (Phase I) II. To assess the impact of the combination of olaparib with durvalumab and tremelimumab on progression free survival (PFS) rates. (Phase II)

SECONDARY OBJECTIVES:

I. To assess the impact of the combination of olaparib with durvalumab and tremelimumab on anti-tumor immune responses in patients with recurrent platinum sensitive or resistant or refractory epithelial ovarian, fallopian tube, or primary peritoneal cancer who carry a germline and/or somatic BRCA1 or BRCA2 mutation and/or a homologous recombination deficiency (HRD).

II. To assess the impact of the combination of olaparib with durvalumab and tremelimumab on PFS and overall survival (OS) in patients with recurrent platinum sensitive or resistant or refractory epithelial ovarian, fallopian tube, or primary peritoneal cancer who carry a germline and/or somatic BRCA1 or BRCA2 mutation and/or a HRD.

OUTLINE: This is a phase I, dose-escalation study of olaparib followed by a phase II study.

Patients receive olaparib orally (PO) twice daily (BID), and tremelimumab intravenously (IV) over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, and every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have platinum-sensitive or platinum-resistant recurrent or persistent or refractory ovarian, fallopian tube, or primary peritoneal carcinoma AND have one or more of the following characteristics documented on a validated platform (documented genetic test report is required). Historic report is permitted.
* A germline BRCA1 or BRCA2 deleterious alteration.
* A somatic mutation in BRCA1 or BRCA2 detected in a tumor sample or on circulating tumor DNA
* Carry a known or likely loss of function alteration in one or more of the homologous recombination or mismatch repair pathways genes
* Demonstrate a genomic phenotype of HR deficiency as measured by a LOH-high score.

  * Recurrent ovarian cancer is defined as recurrence of disease in a patient who achieved initial complete response to primary therapy
  * Persistent ovarian cancer is defined as having residual disease in the form of elevated tumor markers or microscopic or clinically evident disease in a patient who has completed and apparently responded to initial chemotherapy
  * Refractory ovarian cancer is defined as patients who have failed to achieve at least a partial response to therapy including patients with either stable disease or disease progression during primary therapy
  * Platinum-sensitive is defined as achievement of documented response to initial platinum-based treatment and has been off treatment for an extended period of time (more than 6 months)
  * Platinum-resistant is defined as relapse within 6 months of last platinum-based chemotherapy or progression while on platinum-based therapy
* All patients must have measurable disease as defined by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST); measurable disease is defined as 10 mm in the longest diameter by computed tomography (CT) or magnetic resonance imaging (MRI) scan (or no less than double the slice thickness) for non- nodal lesions and >= 15 mm in short axis for nodal lesions, 20 mm by chest X-ray, a lymph node must be >= 15 mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm)
* Must have archival tissue available for PD-L1 assessment
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Patients who have the following risk factors are considered to be at increased risk for cardiac toxicities and may be enrolled only with increased monitoring: i) prior treatment with anthracyclines; ii) prior treatment with trastuzumab; iii) a New York Heart Association classification of II controlled with treatment; iv) prior central thoracic radiation therapy (RT), including RT to the heart
* Any hormonal therapy being taken as a treatment for cancer must be discontinued at least one week prior to registration; continuation of hormone replacement therapy e.g. thyroid hormone replacement therapy is permitted
* Able to tolerate oral medications and no GI illnesses that would preclude absorption of olaparib
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy of > 6 months
* Hemoglobin >= 10 g/dL (no blood transfusion in the 28 days prior to entry [olaparib guidelines])
* White blood cell count (WBC) > 3 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>=1500 per mm^3)
* Platelet count >= 100 x 10^9/L (>= 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN); this will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN
* Creatinine =< 1.5 x ULN, serum creatinine clearance (CL) > 51 ml/min (by the Cockcroft- Gault equation)
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: >= 60 years old and no menses for >=1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1
* Participants of child-bearing potential must agree to use two highly effective and acceptable forms of contraception from screening, throughout their participation in the study and for 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after last dose of durvalumab or olaparib, whichever is the longer time period (e.g., hormonal or barrier method of birth control); should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site); previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 4 weeks (prior use of bevacizumab in the upfront setting is allowed)
* History of discontinuation of any previous treatment with PARP inhibitors, including olaparib, or a PD-1 or PD-L1 inhibitor, including durvalumab or anti-CTLA4 antibody, including tremelimumab due to toxicity.
* Patients with myelodysplastic syndrome/acute myeloid leukemia
* History and/or confirmed interstitial lung disease (ILD)/pneumonitis, extensive bilateral lung disease on high-resolution computed tomography (HRCT) scan
* Concomitant use of a strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, ketoconazole, voriconazole, nefazodone, posaconazole, ritonavir, lopinavir/ritonavir, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) and moderate CYP3A inhibitors (e.g., amprenavir, aprepitant, atazanavir, ciprofloxacin, crizotinib, darunavir/ritonavir, diltiazem, erythromycin, fluconazole. Fosamprenavir, imatinib, verapamil)
* Concomitant use of strong CYP3A inducers (e.g., phenytoin, rifampicin, carbamazepine, St. John's wort) and moderate CYP3A inducers (e.g., bosentan, efavirenz, etravirine, modafinil, nafcillin)
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease (e.g. basal cell or squamous cell carcinoma of the skin)
  * Adequately treated carcinoma in situ without evidence of disease (e.g., breast and cervical cancer in situ)
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, radiotherapy or other investigational agent) =< 21 days prior to the first dose of study drug and within 6 weeks for nitrosourea or mitomycin C)
* Mean QT interval corrected for heart rate (QTcF) >= 470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's correction
* Patients with history of myocardial infarction within 6 months
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity (Common Terminology Criteria for Adverse Events [CTCAE] grade >= 2) from previous anti-cancer therapy; subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
* Any prior grade >= 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > grade 1
* Active or prior documented autoimmune disease within the past 2 years; NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn?s disease, ulcerative colitis)
* Patients with thyroid dysfunction if not adequately controlled
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab, tremelimumab, olaparib or, any excipient
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of, or test positive for, acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab (e.g. live attenuated influenza vaccine [LAIV], measles/mumps/rubella vaccine [MMR], variola virus vaccine [VAR], zoster, yellow fever, etc.)
* Female subjects who are pregnant, breast-feeding, or of reproductive potential who are not employing an effective method of birth control from screening to 180 days after the last dose of durvalumab + tremelimumab + olaparib combination therapy or 90 days after the last dose of durvalumab and olaparib therapy, whichever is the longer time period
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results or, is an unsuitable candidate to receive study drug (e.g. inability to tolerate oral medications which would preclude absorption of olaparib)
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids
* Subjects with uncontrolled seizures
* Dependency on IV hydration or total parenteral nutrition (TPN)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Feinstein Institute for Medical Research/Lennox Hill Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Treatment (Olaparib, Tremelimumab, Durvalumab): Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 300 mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
- Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients: Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 250 mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
  Patients are Platinum Resistant
- Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients: Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 250 mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
  Patients are Platinum Sensitive
Period: Overall Study
Arm/Group | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients
Started | 10 | 20 | 10
Completed | 10 | 20 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients: Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 250 mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Patients are Platinum Sensitive. Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
  Patients are Platinum Resistant
- Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients: Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 250 mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Patients are Platinum Sensitive. Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
  Patients are Platinum Sensitive .
- Total: Total of all reporting groups
Arm/Group | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients | Total
Number analyzed (Participants) | 10 | 20 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 13 | 7 | 25
  >=65 years | 5 | 7 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (6.6) | 61 (10.0) | 60 (10.6) | 61 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 10 | 40
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 19 | 10 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 19 | 10 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicities (DLTs) Defined as the Rate of Drug-related Grade 3-5 Adverse Events Assessed Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (Phase I)
Description: The maximum tolerated dose is defined as the highest dose studied, for which the observed incidence of DLT is less than 33%. Number of Participants with Dose-limiting Toxicities (DLTs) in Phase I and Phase II will be reported.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients: Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 250mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
  Patients are Platinum Resistant
- Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients: Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 250 mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Patients are Platinum Sensitive. Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
  Patients are Platinum Sensitive
Arm/Group | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients
Number analyzed (Participants) | 10 | 20 | 10
Participants | 2 | 0 | 0

2. Primary Outcome: 3 Month Progression Free Survival (PFS) in the All Eligible Patients by Group/Arm
Description: Progression free survival (PFS) rate will be assessed at 3 months in the platinum resistant group using Kaplan-Meier methods. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: At 3 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients
Number analyzed (Participants) | 10 | 20 | 10
Proportion of participants | 0.5 [0.23 to 0.72] | 0.42 [0.24 to 0.60] | 0.88 [0.5 to 0.97]

3. Primary Outcome: 6 Month Progression Free Survival (PFS) in the Platinum Sensitive Group (Phase II)
Description: 6-month progression-free survival rate is the probability of patients remaining alive and progression-free at 6 months from study entry estimated using Kaplan-Meier methods. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesion
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients
Number analyzed (Participants) | 10 | 20 | 10
Proportion of participants | 0.27 [0.07 to 0.52] | 0.21 [0.08 to 0.38] | 0.60 [0.26 to 0.82]

4. Secondary Outcome: Anti-tumor Immune Response of the Treatment Combination Assessed in Tumor Biopsy
Description: Tumor biopsy samples will be examined to evaluate the correlation between clinical activity and the expression level of PD-L1 and tumor-infiltrating lymphocytes changes in biopsies pre and post treatment.
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Treatment (Olaparib, Tremelimumab, Durvalumab)- Platinum Resistant Patients: Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 250mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
  Patients are Platinum Resistant
Arm/Group | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab)- Platinum Resistant Patients | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients
Number analyzed (Participants) | 10 | 20 | 10
Participants
  Immune-related Partial Response (irPR) | 1 | 1 | 1
  Immune-related Stable Disease (irSD) | 4 | 7 | 6
  Immune-related Progressive Disease(irPD) | 4 | 6 | 1
  NE Not Evaluable | 0 | 3 | 2
  Too early | 1 | 3 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS will be summarized and analyzed descriptively via summary frequencies and Kaplan-Meier estimators.
Time Frame: 35 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Treatment I (Olaparib, Tremelimumab, Durvalumab): Durvalumab 1500 mg + Tremelimumab 75 mg + Olaparib 300 mg
  Patients receive olaparib PO BID, and tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment with olaparib continues for up to 12 months in the absence of disease progression or unacceptable toxicity. Treatment with tremelimumab repeats every 4 weeks for up to 4 courses and treatment with durvalumab repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Durvalumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Olaparib: Given PO
  Tremelimumab: Given IV
Arm/Group | Treatment I (Olaparib, Tremelimumab, Durvalumab) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab)- Platinum Resistant Patients | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients
Number analyzed (Participants) | 10 | 20 | 10
Months | 14.9 [4.6 to 34.2] | 9.1 [5.9 to 14.0] | 21.6 [10.8 to NA] — Upper limit of median Overall Survival is not reached

ADVERSE EVENTS:
Time Frame: All-Cause Morality was assessed up to 35 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 8 weeks.
Description: An adverse event or adverse experience (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Therefore, an AE can be ANY unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product.
Arm/Group | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients
All-Cause Mortality (participants affected / at risk) | 8/10 | 15/20 | 4/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 8/20 | 7/10
Other Adverse Events (participants affected / at risk) | 10/10 | 20/20 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) (N=10) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients (N=20) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients (N=10)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Treatment (Olaparib, Tremelimumab, Durvalumab) (N=10) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Resistant Patients (N=20) | Phase II Treatment (Olaparib, Tremelimumab, Durvalumab) - Platinum Sensitive Patients (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (10) | 7 (7) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Adrenal disorder (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Endocrine disorder (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 4 (4) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 6 (10) | 3 (5)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (5) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 7 (8) | 4 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4) | 3 (3)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (9) | 12 (16) | 4 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (4) | 5 (7)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Early satiety (General disorders) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 5 (9) | 7 (7) | 5 (8)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 3 (4) | 0 (0)
Oedema (General disorders) | 2 (3) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Cortisol increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Thyroid function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 4 (4) | 2 (2)
Weight increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 9 (9) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (5) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 2 (4)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (2)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6) | 3 (5)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT02953457/Prot_SAP_000.pdf